CLINICAL TRIAL: NCT05732441
Title: A Randomized Controlled Clinical Trial of a Plant Drug (HuangE Capsule) in the Treatment of Patients With Elevated Psa Prostatitis
Brief Title: Therapeutic Study of Prostatitis With Elevated PSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0354
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2022-07

CONDITIONS: Prostatitis; PSA
MeSH Terms: conditions — Prostatitis

STUDY DESIGN:
Intervention Model Description: 1.Conventional treatment group 2. Conventional treatment group combined with Huange capsule
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment group (No Intervention): Routine treatment protocol are used base on clinical guidelines
- Conventional treatment group combined with Huange capsule (Experimental): Based on the clinical guidelines, the routine treatment was used in addition to Huange Capsule.
  Interventions: Drug: Huange capsule

INTERVENTIONS:
Drug: Huange capsule — Huange Capsule was orally administered (Zhejiang Kangenbe Pharmaceutical Co., Ltd., specification: 0.4g×60 tablets/bottle, GuoYaoZhunZi Z20110006). Administration method: 1.6g each time, three times a day, 40min after breakfast, lunch and dinner. The treatment course was four weeks.
  Arms: Conventional treatment group combined with Huange capsule

SUMMARY:
This clinical study was mainly aimed at exploring the efficacy of herbal medicine (Huange Capsule) in the treatment of patients with prostatitis with elevated PSA.

The main questions it aims to answer are:

1. To evaluate the influence and exact curative effect of huange capsule on serum PSA level of patients with PSA-elevated prostatitis, to improve the specificity of PSA and reduce unnecessary puncture biopsy.
2. To provide evidence-based evidence for clinical efficacy evaluation Subjects will be randomized to a routine regimen with or without the use of Huangge capsules. To evaluate whether the efficacy of the conventional treatment combined with Huange capsule group was superior to that of the conventional medication group.

ELIGIBILITY:
Inclusion Criteria:

1. Compliant with the diagnostic criteria of both Chinese and western medicine for prostatitis;
2. Serum PSA increases, ranging from 4 ng/mL to 10 ng/mL;
3. Male, aged between 18 and 80 years old:
4. B-ultrasound and imaging examination fail to consider the front row cancer;
5. I have not taken any Chinese or western medicine for the treatment of prostatitis in the past two weeks;
6. Those who have signed the informed consent form.

Exclusion Criteria:

1. Patients with frequent micturition caused by combined sexually transmitted diseases and urinary tract infection;
2. oliguria or anuria caused by urinary calculi, prostate cancer, and acute and chronic renal failure;
3. Dysuria caused by neurogenic bladder collapse, bladder neck collapse fibrosis, and urethral stricture;
4. the residual urine volume > 150ml:
5. Losers of invasive treatment of benign prostatic obstruction;
6. Patients with pelvic surgery or injury history that affected the local internal organs, muscles, nerves and other functional states;
7. B-ultrasound shows obvious bladder diverticulum or upper urinary tract obstruction caused by BPH, with impaired renal function;
8. Patients with severe primary diseases such as cardiovascular and cerebrovascular diseases, liver and hematopoietic system, refractory diabetes mellitus, or diabetic neuropathy and psychosis;
9. Patients with serum t-PSA>10ng/ml.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum PSA | 4 weeks
International prostate symptom score | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No